CLINICAL TRIAL: NCT02582580
Title: Effects of Perineal Massage, Vaginal Dilator and Pelvic Floor Muscles Training on the Perineal Integrity Primiparous: A Randomized Controlled Trial Protocol
Brief Title: Effects of Antenatal Pelvic Floor Preparation Techniques for Childbirth
Acronym: EAPFPTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Priscila Godoy Januário Martins Alves, PhD student of the Postgraduate Program in Physical Therapy, Physical Therapy Department, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FAPESP #2015/02244-0; 1.218.385 (Other: Research Ethics Committee)
Record Dates: First submitted 2015-10-14; First posted 2015-10-21 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Pregnancy
Keywords: pelvic floor; perineal trauma; physiotherapy; perineal integrity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Perineal Massage (Active Comparator): Massage is made in the perineum and vagina using your fingers to promote stretching of pelvic floor structures, making them more flexible and distensíveis, avoiding trauma during vaginal birth.
  Interventions: Other: Perineal massage
- Vaginal Dilator (Active Comparator): This device consists of a silicone balloon in an eight shape that, after inserted into the vagina, is inflated by manual pumping, promoting a stretching of the structures around it (hymenal edge, connective tissues and muscles perivaginal). This equipment assists the stretching of tissues around the vagina and the pelvic floor muscles, minimizing the risk of injury from the birth canal during the passage of the baby.
  Interventions: Device: Vaginal Dilator
- Pelvic floor muscles training (Active Comparator): Exercises emphasizing conscious muscle relaxation, i.e., considering a resting time based on the contraction time. The resting time was double of the sustaining time of each contraction up to the 38th week of pregnancy, after remaining fixed this relaxation time up to the moment of delivery. This time was chosen because during the expulsive labor phase, there is a need for the pelvic floor muscles to consciously relax during a long period, in order to facilitate the descendants and rotational movements of the baby's head and consequently, its passage. This exercises does not aim only muscle strength but also contraction promotion, which aims body and perineal awareness, muscle tone, coordination and appropriate motor control to allow an active muscle relaxation in the second labor stage.
  Interventions: Other: Pelvic floor muscles training

INTERVENTIONS:
Other: Perineal massage — Perineal massage should be practiced once a day, from the 34th week of gestation until the beginning of labor. It should obey the following sequence: the pregnant woman must be positioned comfortably and use intimate water based lubricant at her fingertips; start the massage in the outdoor area of the vulva with circular movements of the skin and connective tissue around the vagina and at the central tendon of the perineum, clockwise, clitoris to clitoris; introduce two thumb fingers or index and middle fingers into the vagina at a distance of approximately 4 centimeters; perform internal massaging with laterally semicircles towards the anus for 20 to 30 seconds; put pressure down towards the anus and to each side of the vagina until feeling a slight burning or stretching sensation and hold the position for 2 minutes; massage the lower half of the vaginal introitus in a movement simulating the letter "U". All movements should be repeated four times.
  Other Names: Perineal massage for prevention of perineal trauma
  Arms: Perineal Massage
Device: Vaginal Dilator — Vaginal dilator Epi-No® should be used once a day for 15 minutes, from the 34th week of pregnancy until the beginning of labor. It should be coated with a condom and intimate water based lubricant and then be inserted into the vaginal canal in such way that the balloon stays two centimeters away from the vaginal introitus. The device will be inflated by manual pumping until the tolerable woman's limit. The pregnant woman will be encouraged to daily inflate a greater volume of compressed air into the balloon so that the amount of air is greater than the quantity in the previous day, achieving, day after day, a greater stretching of perivaginal structures, always respecting the individual tolerance limit. The amount of manual pumping imposed to inflate the balloon should be written in an Intervention Diary so that the next use, the pregnant woman will be sure that pumped the device more times than in the previous session.
  Other Names: Epi-No Vaginal Dilator
  Arms: Vaginal Dilator
Other: Pelvic floor muscles training — Pregnant women allocated to this group will perform pelvic floor muscles training. The progression of the protocol of this study will occur gradually in view of the peculiarities that involve the pelvic floor in the gestational stage and the ultimate goal is the promotion of an intact perineum after vaginal delivery. The exercises will obey a sequence, according to the gestation week, considering the following factors/parameters: exercise position, number and sustaining period of slow and fast contractions, and relaxation time between contractions. All contractions should be during the expiratory phase of breathing associated with an isometric contraction of the abdominal muscles and at the end of each series of contractions, perform a one minute interval between sets and in that time perform the diaphragmatic breathing exercise to promote overall relaxation. This protocol should be practiced once a day, every day from the 34th week of gestation until the beginning of labor.
  Other Names: Pelvic floor training for promotion of perineal integrity
  Arms: Pelvic floor muscles training

SUMMARY:
Perineal trauma during childbirth is an important etiological factor of various undesirable complications to women's health, with emphasis on pelvic floor dysfunction. Thus, methods that preserve the perineal integrity have been a challenge to practices among health professionals working in the gravid-puerperal cycle assistance. Despite the remarkable importance of beneficial effects of pelvic floor preparation prior to vaginal birth on prevention of perineal trauma, there are few studies in the literature that point which is the best method to be used to reduce the chances of perineal lesions. Therefore, there is need for more studies to compare existing methods. The objective this present study is to compare the effects of perineal massage, the vaginal dilator and training of the muscles of the pelvic floor to prepare the pelvic floor for vaginal birth on perineal integrity of primiparous. Primigravidae women are selected over 18 years, from the 32th gestational week and wishing to have a vaginal birth. Women will be randomly allocated into 3 groups: perineal massage, vaginal dilator and pelvic floor muscles training and should practice the technique from the 34th week of pregnancy until the time of delivery. All the women will be subject to clinical evaluation, functional assessment of pelvic floor and perineal integrity assessment prior to the beginning of the practice of the technique and between 45 and 60 days after childbirth.

DETAILED DESCRIPTION:
METHODS:

Participants: Primigravidae women over 18 years old will be selected, from the 32th gestational week and wishing to have a vaginal delivery.

Interventions: Pregnant women will be randomly allocated into three groups: perineal massage, vaginal dilator and pelvic floor muscles training. The technique should be practiced from the 34th week of pregnancy until the beginning of labor. Randomization will be done by a researcher who was not involved with the recruitment, assessment and treatment of the participants. All participants will undergo a clinical and functional assessment of the pelvic floor before the beginning of the technique practice, as well as a reassessment of these items and an assessment of perineal integrity between 45 and 60 days after delivery for a blind physiotherapist regarding the interventional procedures.

Objective: To compare the effects of perineal massage, vaginal dilator and pelvic floor muscles training on the perineal integrity of primiparae women.

Outcome: The perineal integrity will be verified by the presence or absence of perineal laceration as well as their characteristics observed immediately after delivery.

Randomization: Participants randomization will be done from a sequence generated by a computer program.

Blinding: The evaluative procedures will be done by a 'blinded' physiotherapist in relation to the intervention procedures and the randomization procedure by a researcher who was not involved with the recruitment, evaluation and participant's treatment.

Discussion: The knowledge of the effects of antenatal pelvic floor preparation techniques on the perineal integrity and pelvic floor muscles function after delivery, will allow a better choice about which approach is the best to pregnant women to prevent perineal trauma.

ELIGIBILITY:
Inclusion Criteria:

* usual risk primigravidae women
* primigravidae women from the 32nd gestational week
* wishing to have a vaginal delivery

Exclusion Criteria:

* pregnant women with pelvic or vaginal surgeries
* presence of pelvic organ prolapse
* intolerance to vaginal palpation
* inability to contract the pelvic floor muscles
* vaginal infections
* neurological and/or cognitive impairments that prevent an understanding of the proposed procedures
* pregnant women who used antenatal pelvic floor methods of preparation prior to study enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Perineal Perineal integrity assessed by the absence or presence of perineal lacerations | This assessment will be done until 60 days after delivery
  Perineal integrity assessed by the absence or presence of perineal lacerations as well as the description of its characteristics: type: classified as single or multiple considering the anterior and posterior perineum region and vaginal wall; Location: classified according to the affected region. Being the anterior region of the perineum, involving the clitoris, left little lip, small right lip, left vestibular region and right vestibular region. The posterior perineum region will be considered when involving left, right and middle region. The vaginal wall will be considered when it presents anterior, back, left back and right back lacerations; Degree of perineal laceration; Laceration form: It will be considered solely for the lacerations affecting posterior perineal region and should be classified as linear, branched and "U" shaped.

SECONDARY OUTCOMES:
Function of the pelvic floor muscles evaluated by the PERFECT method | This assessment will be done at the time of initial evaluation (before the intervention) and between 45 and 60 days after delivery
  Function of the pelvic floor muscles evaluated by the PERFECT method between 45 and 60 days after delivery. This method is a functional assessment of the pelvic floor muscles allowing to analyze the muscle contraction and condition of the fibers. The contraction of pelvic floor muscles will be requested during expiration.

CONTACTS AND LOCATIONS:
Overall Officials: Priscila G Alves, Principal Investigator — Federal University of São Carlos - Physiotherapy Department
Locations (1):
- Federal University of São Carlos - Physical therapy Department, São Carlos, São Paulo, Brazil

REFERENCES:
- [Background] Aasheim V, Nilsen AB, Lukasse M, Reinar LM. Perineal techniques during the second stage of labour for reducing perineal trauma. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD006672. doi: 10.1002/14651858.CD006672.pub2. PMID 22161407
- [Background] Riesco MLG, Costa ASC, Almeida SFS, Basile ALO, Oliveira SMJV. Episiotomia, laceração e integridade perineal em partos normais: análise de fatores associados. Rev. Enferm. UERJ 2011; 19(1): 77-83.
- [Background] Shek KL, Chantarasorn V, Langer S, Phipps H, Dietz HP. Does the Epi-No Birth Trainer reduce levator trauma? A randomised controlled trial. Int Urogynecol J. 2011 Dec;22(12):1521-8. doi: 10.1007/s00192-011-1517-x. Epub 2011 Aug 2. PMID 21809156
- [Background] Beckmann MM, Stock OM. Antenatal perineal massage for reducing perineal trauma. Cochrane Database Syst Rev. 2013 Apr 30;2013(4):CD005123. doi: 10.1002/14651858.CD005123.pub3. PMID 23633325
- [Background] Oliveira LS, Brito LG, Quintana SM, Duarte G, Marcolin AC. Perineal trauma after vaginal delivery in healthy pregnant women. Sao Paulo Med J. 2014;132(4):231-8. doi: 10.1590/1516-3180.2014.1324710. PMID 25055069
- [Background] Kovacs GT, Heath P, Heather C. First Australian trial of the birth-training device Epi-No: a highly significantly increased chance of an intact perineum. Aust N Z J Obstet Gynaecol. 2004 Aug;44(4):347-8. doi: 10.1111/j.1479-828X.2004.00265.x. PMID 15282009
- [Background] Herbert J. Pregnancy and childbirth: the effects on pelvic floor muscles. Nurs Times. 2009 Feb 24-Mar 2;105(7):38-41. PMID 19326654
- [Background] Foroughipour A, Firuzeh F, Ghahiri A, Norbakhsh V, Heidari T. The effect of perineal control with hands-on and hand-poised methods on perineal trauma and delivery outcome. J Res Med Sci. 2011 Aug;16(8):1040-6. PMID 22279480
- [Background] Kopas ML. A review of evidence-based practices for management of the second stage of labor. J Midwifery Womens Health. 2014 May-Jun;59(3):264-76. doi: 10.1111/jmwh.12199. PMID 24850283
- [Background] Zhou F, Wang XD, Li J, Huang GQ, Gao BX. Hyaluronidase for reducing perineal trauma. Cochrane Database Syst Rev. 2014 Feb 5;2014(2):CD010441. doi: 10.1002/14651858.CD010441.pub2. PMID 24497276
- [Background] Brito LG, Ferreira CH, Duarte G, Nogueira AA, Marcolin AC. Antepartum use of Epi-No birth trainer for preventing perineal trauma: systematic review. Int Urogynecol J. 2015 Oct;26(10):1429-36. doi: 10.1007/s00192-015-2687-8. Epub 2015 Apr 8. PMID 25851585
- [Background] Du Y, Xu L, Ding L, Wang Y, Wang Z. The effect of antenatal pelvic floor muscle training on labor and delivery outcomes: a systematic review with meta-analysis. Int Urogynecol J. 2015 Oct;26(10):1415-27. doi: 10.1007/s00192-015-2654-4. Epub 2015 Feb 25. PMID 25711728
- [Background] Salvesen KA, Morkved S. Randomised controlled trial of pelvic floor muscle training during pregnancy. BMJ. 2004 Aug 14;329(7462):378-80. doi: 10.1136/bmj.38163.724306.3A. Epub 2004 Jul 14. PMID 15253920
- [Background] Agur W, Steggles P, Waterfield M, Freeman R. Does antenatal pelvic floor muscle training affect the outcome of labour? A randomised controlled trial. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Jan;19(1):85-8. doi: 10.1007/s00192-007-0391-z. Epub 2007 May 26. PMID 17530154
- [Background] Bo K, Fleten C, Nystad W. Effect of antenatal pelvic floor muscle training on labor and birth. Obstet Gynecol. 2009 Jun;113(6):1279-1284. doi: 10.1097/AOG.0b013e3181a66f40. PMID 19461423
- [Background] Dias LA, Driusso P, Aita DL, Quintana SM, Bo K, Ferreira CH. Effect of pelvic floor muscle training on labour and newborn outcomes: a randomized controlled trial. Rev Bras Fisioter. 2011 Nov-Dec;15(6):487-93. doi: 10.1590/s1413-35552011005000011. Epub 2011 Aug 19. PMID 21860990
- [Background] Bo K, Hilde G, Jensen JS, Siafarikas F, Engh ME. Too tight to give birth? Assessment of pelvic floor muscle function in 277 nulliparous pregnant women. Int Urogynecol J. 2013 Dec;24(12):2065-70. doi: 10.1007/s00192-013-2133-8. Epub 2013 Jun 8. PMID 23749241
- [Background] Boyle R, Hay-Smith EJ, Cody JD, Morkved S. Pelvic floor muscle training for prevention and treatment of urinary and fecal incontinence in antenatal and postnatal women: a short version Cochrane review. Neurourol Urodyn. 2014 Mar;33(3):269-76. doi: 10.1002/nau.22402. Epub 2013 Apr 24. PMID 23616292
- [Background] Dönmez S, Kavlak O. Effects of prenatal perineal massage and Kegel exercises on the integrity of postnatal perine. Health 2015; 7: 495-505.
- [Background] Nagib ABL, Guirro ECO, Palauro VA, Guirro RRJ. Avaliação da sinergia da musculatura abdomino-pélvica em nulíparas com eletromiografia e biofeedback perineal. RBGO 2005; 27(4): 210-5.
- [Background] Laycock J, Jerwood D. Pelvic floor muscle assessment: the PERFECT scheme. Physiotherapy 2001; 87(12): 631-42.
- [Background] Moreira ECH, Brunetto AF, Catanho MM, Nakagawa TH, Yamaguti WPS. Estudo da ação sinérgica dos músculos respiratórios e do assoalho pélvico. Rev Bras Fisioter. 2002; 6(2): 71-6.
- [Background] Labrecque M, Eason E, Marcoux S, Lemieux F, Pinault JJ, Feldman P, Laperriere L. Randomized controlled trial of prevention of perineal trauma by perineal massage during pregnancy. Am J Obstet Gynecol. 1999 Mar;180(3 Pt 1):593-600. doi: 10.1016/s0002-9378(99)70260-7. PMID 10076134
- [Background] Bodner-Adler B, Bodner K, Mayerhofer K. Perineal massage during pregnancy in primiparous women. Int J Gynaecol Obstet. 2002 Jul;78(1):51-3. doi: 10.1016/s0020-7292(02)00065-6. No abstract available. PMID 12113972
- [Background] Kalichman L. Perineal massage to prevent perineal trauma in childbirth. Isr Med Assoc J. 2008 Jul;10(7):531-3. No abstract available. PMID 18751635
- [Background] Jones LE, Marsden N. The application of antenatal perineal massage: a review of literature to determine instruction, dosage and technique. Spring 2008; 102: 8-11.
- [Background] Mei-dan E, Walfisch A, Raz I, Levy A, Hallak M. Perineal massage during pregnancy: a prospective controlled trial. Isr Med Assoc J. 2008 Jul;10(7):499-502. PMID 18751626
- [Background] Hillebrenner J, Wagenpfeil S, Schuchardt R, Schelling M, Schneider KT. [Initial experiences with primiparous women using a new kind of Epi-no labor trainer]. Z Geburtshilfe Neonatol. 2001 Jan-Feb;205(1):12-9. doi: 10.1055/s-2001-14552. German. PMID 11253729
- [Background] Kok J, Tan KH, Koh S, Cheng PS, Lim WY, Yew ML, Yeo GS. Antenatal use of a novel vaginal birth training device by term primiparous women in Singapore. Singapore Med J. 2004 Jul;45(7):318-23. PMID 15221047
- [Background] Ruckhaberle E, Jundt K, Bauerle M, Brisch KH, Ulm K, Dannecker C, Schneider KT. Prospective randomised multicentre trial with the birth trainer EPI-NO for the prevention of perineal trauma. Aust N Z J Obstet Gynaecol. 2009 Oct;49(5):478-83. doi: 10.1111/j.1479-828X.2009.01044.x. PMID 19780729
- [Background] Ashton-Miller JA, Delancey JO. On the biomechanics of vaginal birth and common sequelae. Annu Rev Biomed Eng. 2009;11:163-76. doi: 10.1146/annurev-bioeng-061008-124823. PMID 19591614
- [Background] Ferreira M, Santos P. Princípios da fisiologia do exercício no treino dos músculos do pavimento pélvico. Acta Urológica 2009; 26(3): 31-8.
- [Background] Pereira LC, Botelho S, Marques J, Amorim CF, Lanza AH, Palma P, Riccetto C. Are transversus abdominis/oblique internal and pelvic floor muscles coactivated during pregnancy and postpartum? Neurourol Urodyn. 2013 Jun;32(5):416-9. doi: 10.1002/nau.22315. Epub 2012 Oct 15. PMID 23071085
- [Background] Leite JS. Caracterização das lacerações perineais espontâneas no parto normal. http://www.teses.usp.br/teses/disponiveis/7/7141/tde-20022013-151836/pt-br (2012). Acessado em 08 Jun 2015.
- [Background] Caroci AS, Riesco MLG, Leite JS, Araíjo NM, Scarabotto LB,Oliveira SMJV. Localização das lacerações perineais no parto normal em mulheres primíparas. Rev enferm UERJ 2014; 22(3): 402-8.
- [Background] Cunningham FG. et al. Conduta no trabalho de parto e parto normal. In: Williams Obstetrícia. 20a Ed. Rio de Janeiro: Guanabara Koogan, p. 281-298, 2000.
- [Background] Kettle C, Dowswell T, Ismail KM. Continuous and interrupted suturing techniques for repair of episiotomy or second-degree tears. Cochrane Database Syst Rev. 2012 Nov 14;11(11):CD000947. doi: 10.1002/14651858.CD000947.pub3. PMID 23152204
- [Background] Kettle C, Dowswell T, Ismail KM. Absorbable suture materials for primary repair of episiotomy and second degree tears. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD000006. doi: 10.1002/14651858.CD000006.pub2. PMID 20556745
- [Background] Elharmeel SM, Chaudhary Y, Tan S, Scheermeyer E, Hanafy A, van Driel ML. Surgical repair of spontaneous perineal tears that occur during childbirth versus no intervention. Cochrane Database Syst Rev. 2011 Aug 10;2011(8):CD008534. doi: 10.1002/14651858.CD008534.pub2. PMID 21833968
- [Background] Parente MP, Natal Jorge RM, Mascarenhas T, Silva-Filho AL. The influence of pelvic muscle activation during vaginal delivery. Obstet Gynecol. 2010 Apr;115(4):804-808. doi: 10.1097/AOG.0b013e3181d534cd. PMID 20308842
- [Background] McHugh MP, Cosgrave CH. To stretch or not to stretch: the role of stretching in injury prevention and performance. Scand J Med Sci Sports. 2010 Apr;20(2):169-81. doi: 10.1111/j.1600-0838.2009.01058.x. Epub 2009 Dec 18. PMID 20030776
- [Background] Kruger JA, Dietz HP, Murphy BA. Pelvic floor function in elite nulliparous athletes. Ultrasound Obstet Gynecol. 2007 Jul;30(1):81-5. doi: 10.1002/uog.4027. PMID 17497753